CLINICAL TRIAL: NCT01474304
Title: Intravenous Acetaminophen for Craniotomy Patients: A Single-blinded, Randomized Controlled Trial to Evaluate the Effect of Intravenous Acetaminophen Administered at Induction and Emergence From Craniotomy
Brief Title: Intravenous Acetaminophen for Craniotomy Patients
Acronym: IVAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swedish Medical Center (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IVAC; 20111619 (Other: Western Institutional Review Board (WIRB))
Record Dates: First submitted 2011-11-09; First posted 2011-11-18 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Craniotomy
Keywords: craniotomy; tumor resection; aneurysm; revascularization; opioid; nausea; vomiting; acetaminophen
MeSH Terms: conditions — Aneurysm; Nausea; Vomiting | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Active Comparator): Craniotomy patients will receive a 1000 mg dose of intravenous (IV) acetaminophen before incision and a second 1000 mg dose of IV acetaminophen 6 hours later.
  Interventions: Drug: Acetaminophen
- No acetaminophen (No Intervention): Patients will receive standard of care with no intraoperative doses of acetaminophen.

INTERVENTIONS:
Drug: Acetaminophen — 1000 mg dose intravenous acetaminophen before craniotomy incision and a second 1000 mg dose intravenous acetaminophen 6 hours after surgery
  Arms: Acetaminophen

SUMMARY:
Adding intraoperative IV acetaminophen, in addition to standard analgesics, will decrease opioid requirements over the first 12 hours of postoperative recovery following craniotomy. Opioids exacerbate symptoms of nausea and vomiting. Reducing postoperative opioid use hopefully will reduce incidence of nausea and vomiting in patients after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Weigh at least 50 kg (110.23 lbs)
* Undergoing open, elective intracranial procedure for

  * tumor resection
  * aneurysm clipping
  * revascularization
* Have an ASA (American Society of Anesthesiologists) physical status of 1, 2, 3, or 4
* Able to provide written informed consent

Exclusion Criteria:

* Significant medical disease, laboratory abnormality, or condition that, in the opinion of the investigator, would compromise patient welfare or would otherwise contraindicate study participation
* Unable to communicate symptoms
* Current daily opioid use (>40 mg morphine equivalent)
* Tramadol use
* Treated with MAO (monoamine oxidase inhibitors) inhibitors within 10 days of surgery
* Treated with any amount of acetaminophen within 8 hours of anesthesia for surgery
* Allergic or hypersensitive to acetaminophen or any contraindications per manufacturer's guidelines
* Pregnancy
* Impaired liver function
* Participation in interventional clinical study within the last 30 days
* Known or suspected history of alcohol or drug abuse
* Surgery for resection of acoustic neuroma
* Transphenoidal tumor resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Total narcotic dose administered over the first 12 hours of postoperative recovery. | 12 hours
  Intensive care nurses will ask subject about pain and nausea every 15 minutes for the first two hours immediately after surgery and then every hour afterward for up to 12 hours. Nurses will record subject response and opioid doses given.

SECONDARY OUTCOMES:
Incidence of nausea during postoperative recovery | 12 hours
Incidence of vomiting during postoperative recovery | 12 hours
Severity of nausea during postoperative recovery | 12 hours
Severity of vomiting during postoperative recovery | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Lam, MD, FRCPC, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center Cherry Hill Campus, Seattle, Washington, United States